CLINICAL TRIAL: NCT05429203
Title: Comparison of Outcomes in Patients Undergoing Endoscopic Retrograde Cholangiopancreatoscopy (ERCP) Using Duodenoscope With Single-use Distal Cover and Conventional Reusable Duodenoscope: A Randomized Controlled Trial
Brief Title: Comparison of Duodenoscope With Single-use Distal Cover and the Conventional Reusable Duodenoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Subhas Banerjee, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 65189
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Biliary Disease; Pancreatic Disease; Choledocholithiasis; Biliary Obstruction; Biliary Tract Neoplasms; Pancreatic Neoplasms
Keywords: ERCP; Duodenoscope; Duodenoscope with single-use distal cover
MeSH Terms: conditions — Gallbladder Diseases; Pancreatic Diseases; Choledocholithiasis; Biliary Tract Neoplasms; Pancreatic Neoplasms | interventions — Duodenoscopes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Duodenoscope with single-use distal cover (Active Comparator): Patients will undergo ERCP using a duodenoscope with a single-use distal cover
  Interventions: Device: Duodenoscope with single-use distal cover
- Conventional Duodenoscope (Active Comparator): Patients will undergo ERCP using a conventional duodenoscope
  Interventions: Device: Conventional duodenoscope

INTERVENTIONS:
Device: Duodenoscope with single-use distal cover — Newer duodenoscope with a single-use distal cover
  Arms: Duodenoscope with single-use distal cover
Device: Conventional duodenoscope — Conventional duodenoscope with standard methods of reprocessing
  Arms: Conventional Duodenoscope

SUMMARY:
The purpose of the study is to compare the success rates of procedure success and complication rates in patients undergoing Endoscopic retrograde cholangiopancreatography (ERCP) using two types of currently available endoscopes. These are (1) duodenoscope with a Single-use distal cover or (2) a conventional reusable duodenoscope.

DETAILED DESCRIPTION:
The risks associated with the ERCP procedure will be explained to patients who meets the eligibility criteria. Consenting patients will be randomized to undergo Endoscopic retrograde cholangiopancreatography (ERCP) using either (1) a duodenoscope with a Single-use distal cover or (2) a conventional reusable duodenoscope. Assessments will be made during, and immediately after the procedure, then patients will be called after 1 week, 1 month, and 3 months after the procedure to get information about adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ERCP for biliary and pancreatic conditions
* Age > 18 years old

Exclusion Criteria:

* Vulnerable patient groups including pregnant women
* Patients who are unable to consent
* Patients with known cholangitis
* Patients with known Carbapenem-Resistant Enterobacteriaceae (CRE) or any other multi-drug resistant organisms (MDRO) infection
* Surgically altered anatomy except for Billroth I

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subhas Banerjee, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bang JY, Rosch T, Kim HM, Thakkar S, Robalino Gonzaga E, Tharian B, Inamdar S, Lee LS, Yachimski P, Jamidar P, Muniraj T, DiMaio C, Kumta N, Sethi A, Draganov P, Yang D, Seoud T, Perisetti A, Bondi G, Kirtane S, Hawes R, Wilcox CM, Kozarek R, Reddy DN, Varadarajulu S. Prospective evaluation of an assessment tool for technical performance of duodenoscopes. Dig Endosc. 2021 Jul;33(5):822-828. doi: 10.1111/den.13856. Epub 2020 Nov 17. PMID 33007136

RESULTS

PARTICIPANT FLOW:
Groups:
- Duodenoscope With Disposable Distal End Caps: Patients will undergo endoscopic retrograde cholangiopancreatography (ERCP) using a duodenoscope with a single-use distal cover.
- Conventional Reusable Duodenoscope: Patients will undergo ERCP using a conventional duodenoscope.
Period: Overall Study
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Started | 159 | 160
Completed | 159 | 160
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Duodenoscope With Disposable Distal End Caps: Patients will undergo ERCP using a duodenoscope with a single-use distal cover.
- Total: Total of all reporting groups
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope | Total
Number analyzed (Participants) | 159 | 160 | 319
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.5 [48 to 72.7] | 65 [52 to 72.5] | 65 [50 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 74 | 130
  Male | 103 | 86 | 189
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 41 | 48 | 89
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 33 | 60
  White | 75 | 62 | 137
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 17 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 159 | 160 | 319
Previous ERCP [Count of Participants; unit: Participants] — Index: Patients having ERCP for the first time. Repeat: Patient who had prior ERCP.
  Participants
    Index | 45 | 44 | 89
    Repeat | 114 | 116 | 230

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedure-related Adverse Events
Description: Patients undergoing Endoscopic retrograde cholangiopancreatography (ERCP) using either of the 2 duodenoscopes were assessed for superficial mucosal injury, perforation of the stomach or intestine, mucosal bleeding, pancreatitis, infection, death or any other symptom reported by the patient.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Number analyzed (Participants) | 159 | 160
Participants | 8 | 9
Statistical Analysis 1: Comparison: Duodenoscope With Disposable Distal End Caps vs Conventional Reusable Duodenoscope; Test type: Other; p = 0.8, Chi-squared — The a priori threshold for statistical significance was <0.05

2. Secondary Outcome: Duodenoscope Maneuverability: Intubation Into Esophagus
Description: Providers assessed the 2 duodenoscopes for maneuverability during the procedure in patients undergoing ERCP, using a previously defined scoring system which uses a 5-point scale ranging from 1 to 5, with 1 being easy to perform, 2 minimal difficulty, 3 moderate difficulty, 4 severe difficulty and 5 unable to complete the requisite maneuver.
Time Frame: Maneuverability will be assessed only during the procedure (approximately 10 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Number analyzed (Participants) | 159 | 160
Participants
  Rating = 1 | 153 | 154
  Rating = 2 | 5 | 5
  Rating = 3 | 1 | 1
  Rating = 4 | 0 | 0
  Rating = 5 | 0 | 0
Statistical Analysis 1: Comparison: Duodenoscope With Disposable Distal End Caps vs Conventional Reusable Duodenoscope; Test type: Other; p = 1, Fisher Exact — The a priori threshold for statistical significance was <0.05

3. Secondary Outcome: Duodenoscope Maneuverability: Passage Into Stomach
Description: as for outcome 2
Time Frame: Maneuverability will be assessed only during the procedure (approximately 10 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Number analyzed (Participants) | 159 | 160
Participants
  Rating = 1 | 153 | 155
  Rating = 2 | 3 | 2
  Rating = 3 | 3 | 2
  Rating = 4 | 0 | 1
  Rating = 5 | 0 | 0
Statistical Analysis 1: Comparison: Duodenoscope With Disposable Distal End Caps vs Conventional Reusable Duodenoscope; Test type: Other; p = 0.7, Fisher Exact — The a priori threshold for statistical significance was <0.05

4. Secondary Outcome: Duodenoscope Maneuverability: Navigation Across Pylorus
Description: as for outcome 2
Time Frame: Maneuverability will be assessed only during the procedure (approximately 10 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Number analyzed (Participants) | 159 | 160
Participants
  Rating = 1 | 151 | 155
  Rating = 2 | 3 | 4
  Rating = 3 | 1 | 1
  Rating = 4 | 2 | 0
  Rating = 5 | 2 | 0
Statistical Analysis 1: Comparison: Duodenoscope With Disposable Distal End Caps vs Conventional Reusable Duodenoscope; Test type: Other; p = 0.4, Fisher Exact — The a priori threshold for statistical significance was <0.05

5. Secondary Outcome: Duodenoscope Maneuverability: Achieving Short Position of the Scope
Description: as for outcome 2
Time Frame: Maneuverability will be assessed only during the procedure (approximately 10 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Number analyzed (Participants) | 159 | 160
Participants
  Rating = 1 | 154 | 155
  Rating = 2 | 3 | 4
  Rating = 3 | 2 | 1
  Rating = 4 | 0 | 0
  Rating = 5 | 0 | 0
Statistical Analysis 1: Comparison: Duodenoscope With Disposable Distal End Caps vs Conventional Reusable Duodenoscope; Test type: Other; p = 0.8, Fisher Exact — The a priori threshold for statistical significance was <0.05

6. Secondary Outcome: Duodenoscope Maneuverability: Achieving Optimal Papillary Position
Description: as for outcome 2
Time Frame: Maneuverability will be assessed only during the procedure (approximately 10 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Number analyzed (Participants) | 159 | 160
Participants
  Rating = 1 | 154 | 154
  Rating = 2 | 4 | 4
  Rating = 3 | 1 | 2
  Rating = 4 | 0 | 0
  Rating = 5 | 0 | 0
Statistical Analysis 1: Comparison: Duodenoscope With Disposable Distal End Caps vs Conventional Reusable Duodenoscope; Test type: Other; p = 0.8, Fisher Exact — The a priori threshold for statistical significance was <0.05

7. Secondary Outcome: Duodenoscope Mechanical Characteristics Profile: Scope Stiffness
Description: Providers assessed the 2 duodenoscopes for their mechanical characteristics during the procedure in patients undergoing ERCP. Each characteristic was assessed using a published 5-point scoring system, with 1 being easy to perform, 2 minimal difficulty, 3 moderate difficulty, 4 severe difficulty and 5 unable to complete the requisite maneuver.
Time Frame: Mechanical characteristics assessed only during the procedure (approximately 15 minutes)
Measure: Count of Participants; unit: Participants
Groups:
- Duodenoscope With Disposable Distal End Caps: Patients underwent endoscopic retrograde cholangiopancreatography (ERCP) using a duodenoscope with a single-use distal cover.
- Conventional Reusable Duodenoscope: Patients underwent ERCP using a conventional duodenoscope.
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Number analyzed (Participants) | 159 | 160
Participants
  Rating = 1 | 155 | 155
  Rating = 2 | 4 | 5
  Rating = 3 | 0 | 0
  Rating = 4 | 0 | 0
  Rating = 5 | 0 | 0
Statistical Analysis 1: Comparison: Duodenoscope With Disposable Distal End Caps vs Conventional Reusable Duodenoscope; Test type: Other; p = 0.7, Fisher Exact — The a priori threshold for statistical significance was <0.05

8. Secondary Outcome: Duodenoscope Mechanical Characteristics Profile: Air-water Button Functionality
Description: Providers assessed the 2 duodenoscopes for their mechanical characteristics during the procedure in patients undergoing ERCP. Each characteristic was assessed using a published 5-point scoring system, with 1 being no water leakage or no difficulty in applying suction or inflating air, 2 minimal leakage or minimal difficulty with suction or inflation, 3 moderate leakage or difficulty, 4 severe leakage or difficulty and 5 unable to perform the requisite function.
Time Frame: Mechanical characteristics assessed only during the procedure (approximately 15 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Number analyzed (Participants) | 159 | 160
Participants
  Rating = 1 | 155 | 156
  Rating = 2 | 3 | 4
  Rating = 3 | 1 | 0
  Rating = 4 | 0 | 0
  Rating = 5 | 0 | 0
Statistical Analysis 1: Comparison: Duodenoscope With Disposable Distal End Caps vs Conventional Reusable Duodenoscope; Test type: Other; p = 0.6, Fisher Exact — The a priori threshold for statistical significance was <0.05

9. Secondary Outcome: Duodenoscope Mechanical Characteristics Profile: Elevator Efficiency
Description: as for outcome 7
Time Frame: Mechanical characteristics assessed only during the procedure (approximately 15 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Number analyzed (Participants) | 159 | 160
Participants
  Rating = 1 | 157 | 158
  Rating = 2 | 1 | 2
  Rating = 3 | 1 | 0
  Rating = 4 | 0 | 0
  Rating = 5 | 0 | 0
Statistical Analysis 1: Comparison: Duodenoscope With Disposable Distal End Caps vs Conventional Reusable Duodenoscope; Test type: Other; p = 0.5, Fisher Exact — The a priori threshold for statistical significance was <0.05

10. Secondary Outcome: Duodenoscope Mechanical Characteristics Profile: Hand Strain
Description: Providers assessed the 2 duodenoscopes for their mechanical characteristics during the procedure in patients undergoing ERCP. Each characteristic was assessed using a published 5-point scoring system, with 1 being no strain, 2 minimal strain, 3 moderate strain, 4 severe strain and 5 unable to complete the procedure.
Time Frame: Mechanical characteristics assessed only during the procedure (approximately 15 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Number analyzed (Participants) | 159 | 160
Participants
  Rating = 1 | 157 | 158
  Rating = 2 | 2 | 2
  Rating = 3 | 0 | 0
  Rating = 4 | 0 | 0
  Rating = 5 | 0 | 0
Statistical Analysis 1: Comparison: Duodenoscope With Disposable Distal End Caps vs Conventional Reusable Duodenoscope; Test type: Other; p = 0.9, Fisher Exact — The a priori threshold for statistical significance was <0.05

11. Secondary Outcome: Duodenoscope Imaging Characteristics Profile: Image Quality
Description: Providers assessed the 2 duodenoscopes for their imaging characteristics during the procedure in patients undergoing ERCP. Each characteristic was assessed using a published 5-point scoring system, with 1 being superior, 2 good, 3 satisfactory, 4 suboptimal and 5 unable to visualize or achieve stability of image resulting in termination of procedure.
Time Frame: Imaging characteristics were assessed only during the procedure (approximately 15 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Number analyzed (Participants) | 159 | 160
Participants
  Rating = 1 | 154 | 154
  Rating = 2 | 4 | 4
  Rating = 3 | 1 | 2
  Rating = 4 | 0 | 0
  Rating = 5 | 0 | 0
Statistical Analysis 1: Comparison: Duodenoscope With Disposable Distal End Caps vs Conventional Reusable Duodenoscope; Test type: Other; p = 0.8, Fisher Exact — The a priori threshold for statistical significance was <0.05

12. Secondary Outcome: Duodenoscope Imaging Characteristics Profile: Image Stability
Description: as for outcome 11
Time Frame: Imaging characteristics were assessed only during the procedure (approximately 15 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Number analyzed (Participants) | 159 | 160
Participants
  Rating = 1 | 156 | 157
  Rating = 2 | 3 | 3
  Rating = 3 | 0 | 0
  Rating = 4 | 0 | 0
  Rating = 5 | 0 | 0
Statistical Analysis 1: Comparison: Duodenoscope With Disposable Distal End Caps vs Conventional Reusable Duodenoscope; Test type: Other; p = 0.9, Fisher Exact — the a priori threshold for statistical significance was <0.05

13. Secondary Outcome: Number of Participant With Procure Success (Ability to Perform Interventions)
Description: Patients undergoing Endoscopic retrograde cholangiopancreatography (ERCP) using either of the 2 duodenoscopes will be assessed for their ability to perform endoscopic maneuvers like sphincterotomy, balloon sweep, use of basket/mechanical lithotriptor, stone clearance, stricture dilation using balloon/catheter, stent insertion, stent removal and use of single operator cholangioscopy/pancreatoscopy.
Time Frame: 30-60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
Number analyzed (Participants) | 159 | 160
Participants | 154 | 155

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Duodenoscope With Disposable Distal End Caps | Conventional Reusable Duodenoscope
All-Cause Mortality (participants affected / at risk) | 1/159 | 0/160
Serious Adverse Events (participants affected / at risk) | 8/159 | 9/160
Other Adverse Events (participants affected / at risk) | 8/159 | 8/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duodenoscope With Disposable Distal End Caps (N=159) | Conventional Reusable Duodenoscope (N=160)
Post ERCP pancreatitis (PEP) (Gastrointestinal disorders) | 6 | 5
Post-sphincterotomy bleeding (Surgical and medical procedures) | 1 | 3
Cholangitis (Hepatobiliary disorders) | 1 | 1
Perforation (Surgical and medical procedures) | 1 | 1
Liver failure (Hepatobiliary disorders) | 1 | 0 — Unrelated to treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Duodenoscope With Disposable Distal End Caps (N=159) | Conventional Reusable Duodenoscope (N=160)
Abdomen pain (without post-ERCP pancreatitis) (Gastrointestinal disorders) | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT05429203/Prot_SAP_000.pdf